CLINICAL TRIAL: NCT01943240
Title: Improvement of Analgesia With Addition of Pectoral Nerve Block to Thoracic Paravertebral Blocks in Unilateral Total Simple Mastectomy
Brief Title: Pectoral Nerve Blockade in Mastectomy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient population of eligible patients; none enrolled
Sponsor: Timothy R Petersen (Other)
Responsible Party: Sponsor-Investigator, Timothy R Petersen, Research Information Specialist, University of New Mexico
Organization: University of New Mexico (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pec block
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Postoperative Pain; Breast Cancer
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Paravertebral peripheral nerve blockade with with 4 mL of 0.5% ropivacaine at each of six levels, plus 10 cc of 0.375% ropivacaine for pectoral nerve block
  Interventions: Drug: Paravertebral nerve block: 4 mL ropivacaine 0.5% at each of six levels; Drug: 10 cc of 0.375% ropivacaine pectoral nerve block
- Group S (Active Comparator): Paravertebral peripheral nerve blockade with 4 mL of 0.5% ropivacaine at each of six levels, plus 10 cc of normal saline for pectoral nerve block.
  Interventions: Drug: Paravertebral nerve block: 4 mL ropivacaine 0.5% at each of six levels

INTERVENTIONS:
Drug: Paravertebral nerve block: 4 mL ropivacaine 0.5% at each of six levels
Drug: 10 cc of 0.375% ropivacaine pectoral nerve block
  Arms: Group A

SUMMARY:
Our routine practice for patients undergoing mastectomy is to include paravertebral peripheral nerve blockade for postoperative analgesia. This study investigates whether the addition of another nerve block targeting the pectoral nerves will improve that analgesia.

DETAILED DESCRIPTION:
Randomization:

20 patients will be randomized into 2 groups. Both groups will receive paravertebral blocks with 4 mL of 0.5% ropivacaine at each of six levels.

Group A: Active group with 10 cc of 0.375% ropivacaine (16) pectoral nerve block Group S: Placebo group with 10 cc of normal saline for pectoral nerve block

Blinding:

The injectate contents for the lateral pectoral nerve block will be blinded to all personnel involved in performing the block, all personnel involved in the general anesthesia and all personnel involved in assessing the patient for pain in the postoperative recovery period.

Procedure:

All study patients will be consented for a paravertebral block and a lateral pectoral nerve block as per institutional standards. Pre-block procedure will follow the standard operating procedures of the institution including time out, intravenous access, oxygen supplementation, electrocardiogram, pulse oximeter and automated noninvasive blood pressure monitoring.

Paravertebral block will be performed as usual, as described by Moller (17). Patients will be in a sitting position with a staff member standing in front of the patient to ensure safety. The surgical site will be marked both in the front and on the back of the patient with dual confirmation from the consent and the patient. Mild sedation will be given using midazolam 2 mg and fentanyl 100 µg. The superior aspects of the spinous processes of thoracic levels C7-T5 will be identified with palpation. The needle entry site will be marked at 2.5 cm lateral to each spinous process ipsilateral to the operative breast. Using a 22-gauge, Tuohy needle (B Braun Medical Inc, Bethlehem, PA, USA) attached via extension tubing to a syringe, the needle will be advanced anteriorly in the parasagittal plane (perpendicular to the back in all directions) until it contacts the transverse process. The needle will then be withdrawn to the subcutaneous tissue and angled to walk off the caudal edge of the transverse process. From the caudal edge, it will then be advanced anteriorly approximately 1 cm. (17) After negative aspiration of the syringe, 4 mL of 0.5% ropivacaine will be injected at each of the six levels. These injections correspond to the T1-T6 spinal root levels.

The lateral pectoral nerve block is performed as described by Blanco (15). A linear ultrasound probe (L28 sonosite, Seattle, WA, USA) will be placed in a sagittal paramedian fashion inferior to the lateral third of the ipsilateral clavicle medial to the coracoid. Once the pectoralis major muscle and axillary artery is identified, the thoraco-acromial artery is identified between the pectoralis major and pectoralis minor muscle and confirmed with color Doppler. The lateral pectoral nerve is consistently located adjacent to the artery. (15) Ten mL of study injectate (16) will be delivered using an in-plane technique via a 80 mm echogenic (Pajunk, Germany) needle adjacent to the artery and into the inter-pectoral plane. Care is taken to avoid intramuscular and intravascular injection. The contents of the injectate will be blinded to any personnel involved in performing the block, general anesthesia, or post operative care.

All patients will proceed with general anesthesia. Induction will be with propofol and maintenance with desflurane. Airway management will be with an LMA without use of muscle relaxant as per standard practice. Fentanyl will be used intraoperatively to treat pain. Hydromorphone will be used to treat pain in the post- operative setting. No NSAID or acetaminophen will be given in any route. For prevention of post operative nausea and vomiting, all patients will be given a 1.5mg scopolamine patch, 8 mg of dexamethasone at the beginning of surgery,(18) and 4 mg of ondansetron at closing.

Any supplemental local anesthetic infiltration by surgeons will be noted.

Assessment:

Standard post anesthetic care unit assessment (PACU) of numerical rating pain scale score will be performed as per standard protocol. Hydromorphone will be used to treat pain in the post-operative setting. If pain control is inadequate, other analgesics may be prescribed at the discretion of anesthesia providers involved in the case as per standard practice. Additional anti-emetics may be prescribed and used whenever necessary.

Data collection includes total preoperative, intraoperative fentanyl and total post- operative hydromorphone. Data collection concludes when the patient has met PACU discharge criteria or 2 hours after arousal, whichever is sooner. Time of PACU admission and when the patient has met PACU discharge criteria is recorded. Any supplementary local anesthetics or analgesia will also be noted. Prior to PACU discharge, a blinded assessor will assess the patient for any reduced sensation to cold in the distribution of the radial, ulnar, median nerves in the hand and musculocutaneous nerve in the arm as well as the motor integrity of the 4 said nerves. Patient grip strength will be measured on the surgical and contralateral sides with a grip dynamometer. Three iterations of measurements will be taken prior to the nerve block procedure and again when the patient is ready for discharge from PACU.

Patient satisfaction will be assessed at PACU discharge with a standard question, "Thinking about your nerve blocks, how satisfied were you with them: where 1 is not at all, 4 is in the middle, and 7 is completely satisfied?" scored on a 7-point Likert scale.

Any complications will be noted, with follow up and management as per the institution standard operating procedure. Known risks of regional anesthesia include small risks of infection, swelling and bleeding, and extremely rare risks of nerve damage, collapsed lung, seizure, and death. Unanticipated adverse events will also be reported to the PI for evaluation and possible reporting to the HRRC, according to HRRC policy.

Statistical analysis:

Demonstrating that non-blocked patients' analgesic requirements differ from the hypothesized mean for blocked patients at α=0.05 and 80% power will require a total sample size of 16 (8/group). This estimate is based on observational data for non-blocked patients from our own practice, and our estimate of the minimum clinically-significant difference in analgesic requirements to be expected in blocked patients. We currently estimate that enrollment of 20 participants should be sufficient to accumulate 16 who complete the protocol , and will apply to HRRC for an amendment to enroll more should that be necessary.

Statistical analysis of most outcomes (opioid consumption, pain score, time to discharge) will be carried out with Wilcoxon tests or t-tests, as appropriate. The remaining outcomes (PONV incidence, incidence of weakness or modified sensation in ipsilateral upper limb) will be analyzed with proportion tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Able to provide own consent
* Simple mastectomy at University of New Mexico Hospital without planned axillary surgery

Exclusion Criteria:

* Spinal deformity or pathology
* Chest wall deformity or pathology
* BMI >40
* Bilateral simple mastectomy
* Refusal of regional anesthesia
* Chronic pain
* History of recent drug or alcohol abuse
* History of recent psychiatric problems
* Allergies to lidocaine or ropivacaine
* Allergies to fentanyl or hydromorphone
* Surgery that extends beyond the original plan to include axillary exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption in post anesthesia care unit (PACU) | Up to 8 hours

SECONDARY OUTCOMES:
Maximum pain score in PACU (numerical rating scale) | Up to 8 hours
Time to meet PACU discharge criteria | Up to 8 hours
Patient satisfaction with block | 1 day
Postoperative nausea and vomiting (PONV) | Up to 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Lam, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States